CLINICAL TRIAL: NCT02497859
Title: Does Higher Protein Quality Breakfast Reduce Energy Intake When Following a Weight Loss Diet Plan?
Brief Title: Breakfast Intake and Satiety Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Nikhil Dhurandhar, Professor, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 505159
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Weight Reduction; Weight Loss Diet; Satiety Response; Insulin; Glucagon-Like Peptide 1; PYY (3-36) peptide; Ghrelin; Glucose; Eggs; Protein; Energy Intake; Breakfast
MeSH Terms: conditions — Obesity; Weight Loss; Insulin Resistance | interventions — Diet, Reducing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egg Breakfast (EB) (Experimental): The EB will receive the following breakfast:
  2 scrambled eggs, 120 mL skim milk, 2 slices of Mrs. Bairds® Extra Thin White Bread, 5 g of butter, and 18 g of Smuckers® Strawberry Jam.
  Interventions: Behavioral: Egg Breakfast (EB); Behavioral: Weight Loss Counseling; Behavioral: Weight Loss Diet
- Cereal Breakfast (CB) (Active Comparator): The CB will receive the following breakfast:
  1.5 cups of Special K® Ready-to-Eat Original Cereal, 200 ml Silk® Original Soymilk, 1 slice of Nature's Own® Double Fiber Wheat Bread, 13 g of butter, and 10 g of Smuckers® Sugar-Free Strawberry Jam.
  Interventions: Behavioral: Cereal Breakfast (CB); Behavioral: Weight Loss Counseling; Behavioral: Weight Loss Diet

INTERVENTIONS:
Behavioral: Egg Breakfast (EB) — The EB will receive a breakfast of higher quality protein, but similar in macronutrient and energy density than the active comparator. The EB will have the following energy density, macronutrient composition, and protein score: weight 291 g,energy 400 kcal, energy density 1.37 kcal/g, carbohydrate 42.9%, fat 35.5%, protein 19.8%, protein digestibility corrected amino acid score (PDCAAS) 100, leucine 1.77 g, glycemic load 24, fiber 1.0 g.
  Arms: Egg Breakfast (EB)
Behavioral: Cereal Breakfast (CB) — The CB will receive a breakfast of lower quality protein, but similar in macronutrient and energy density than the experimental treatment. The CB will have the following energy density, macronutrient composition, and protein score: weight 293 g, energy 398 kcal, energy density 1.3 kcal/g, carbohydrate 44.8%, fat 35.4%, protein 19.8%, protein digestibility corrected amino acid score (PDCAAS) 42, leucine 0.48 g, glycemic load 30.8, fiber 4.4 g.
  Arms: Cereal Breakfast (CB)
Behavioral: Weight Loss Counseling — Weight loss counseling will be administered by a Registered Dietitian and will utilize information and materials derived from the Evidence Analysis Library (EAL) of the Academy of Nutrition and Dietetics (AND). Topics including portion control, macronutrient distribution, snacking, eating out, cooking and grocery shopping, will be discussed. Self-monitoring, motivational interviewing, goal setting, and problem solving will be the behavioral strategies used during counseling.
Behavioral: Weight Loss Diet — Energy intake for study duration will be prescribed at 1,200-1,500 kcals adjusted for each individual's body weight.

SUMMARY:
The experiments in this study will assess if while following a reduced energy diet, eating a breakfast with higher protein quality will enhance weight loss compared to another breakfast with lower protein quality, but matched for energy density and macronutrient composition.

DETAILED DESCRIPTION:
There will be 2 experiments in this pilot study. Both will be randomized crossover study designs with subjects beginning on either an egg breakfast of higher protein quality or cereal breakfast of lower protein quality, and reversing to receive the breakfast not previously ingested. The subjects will consume breakfasts under supervision at our clinic on all days of the study, except for weekends. Subjects will be advised to continue eating their breakfast at home on weekends. All subjects will receive weight loss counseling and follow a weight loss diet for 2 weeks. Experiment 1 will test the hypothesis that when on a reduced calorie diet, intake of an egg breakfast compared to cereal breakfast increases satiety, reduces lunch time energy consumption and reduces dinner time energy consumption in clinical and free living condition. Insulin, glucagon-like peptide-1, peptide YY 3-36, ghrelin, plasma glucose, baseline and post intervention anthropomorphic measurements, and hunger questionnaires completed during the consumption of both breakfasts and subsequent meals will be compared. Experiment 2 will compare the effects of the two breakfasts on intake of foods considered tempting or highly palatable, and assessment of energy intake pre/post test lunch followed by offering brownies. It is hypothesized that consumption of an egg breakfast compared to cereal breakfast, will help in reducing intake of foods considered tempting.

ELIGIBILITY:
Inclusion Criteria:

* Calculated BMI of 25.0-39.9 kg/m2
* Sedentary (< 3 hours/week of moderate intensity physical activity)
* Otherwise healthy

Exclusion Criteria:

* ≥5% body weight loss or gain in the three months preceding the study
* Post-menopausal (has not had period for 12 months)
* Plans to begin an exercise program or change current exercise routines between initiation of study and final study
* Anyone following a medical diet prescription
* Anyone with a chronic disease including type II diabetes, hypothyroidism, hypoparathyroidism, cardiovascular disease, cancer of any type
* Health conditions and chronic illness that contraindicate behavioral weight loss treatment using a low calorie diet
* Anyone who is currently pregnant, or lactating
* Medications that may influence or inhibit appetite, sensory functioning, or hormone signaling
* Plans to begin taking any supplements that may influence weight loss
* Report of medical condition or surgical intervention that affects swallowing or chewing ability
* Anyone with a pacemaker or other internal medical device
* Any practicing vegans or vegetarians
* Any practicing gluten-free diet
* Allergy, aversion, or dislike to any of the foods offered for meals

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in subjective hunger questionnaire (Visual Analog Scale) | Change in scores (arbitrary units AU) from 30 minutes prior to breakfast consumption to 240 minutes post consumption.
Change in serum satiety and hunger hormones | Change (AU) from 30 minutes prior to breakfast consumption to 240 minutes post consumption.
  Concentrations of ghrelin, GLP1, PYY 3-36, insulin, and serum glucose will be determined. This is only for experiment 1.
Energy intake (kcal) during ad libitum lunch | Test day 7 (30 minutes for buffet).
  This is for experiment 1.
Energy intake (kcal) during ad libitum lunch | Test day 14 (30 minutes for buffet).
  This is for experiment 1.
Energy intake (kcal) during ad libitum dinner | Test day 7 (30 minutes for buffet).
  This is for experiment 1.
Energy intake (kcal) during ad libitum dinner | Test day 14 (30 minutes for buffet).
  This is for experiment 1.
Energy intake (kcal) during ad libitum lunch | Test day 7 (30 minutes for buffet).
  This is for experiment 2. Chocolate brownies will be added to the test lunch.
Energy intake (kcal) during ad libitum lunch | Test day 14 (30 minutes for buffet).
  This is for experiment 2. Chocolate brownies will be added to the test lunch.

SECONDARY OUTCOMES:
Change in body weight in kilograms | Change in kilograms from baseline to test day 7.
Change in body weight in kilograms | Change in kilograms from test day 7 to test day 14.
Change in waist and hip circumference in centimeters | Change in centimeters from baseline to test day 7.
Change in waist and hip circumference in centimeters | Change in centimeters from test day 7 to test day 14.
Change in blood pressure (mm Hg) | Change in mm Hg from baseline to test day 7.
Change in blood pressure (mm Hg) | Change in mm Hg from test day 7 to test day 14.
Change in fat mass and lean body mass percentage | Change in percentage from test day 0 to test day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Dhurandhar, PhD, Principal Investigator — Chair of the Nutritional Sciences Department
Locations (1):
- Texas Tech University - Department of Nutritional Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayham BE, Greenway FL, Johnson WD, Dhurandhar NV. A randomized trial to manipulate the quality instead of quantity of dietary proteins to influence the markers of satiety. J Diabetes Complications. 2014 Jul-Aug;28(4):547-52. doi: 10.1016/j.jdiacomp.2014.02.002. Epub 2014 Feb 13. PMID 24703415
- [Background] Vander Wal JS, Gupta A, Khosla P, Dhurandhar NV. Egg breakfast enhances weight loss. Int J Obes (Lond). 2008 Oct;32(10):1545-51. doi: 10.1038/ijo.2008.130. Epub 2008 Aug 5. PMID 18679412
- [Background] Vander Wal JS, Marth JM, Khosla P, Jen KL, Dhurandhar NV. Short-term effect of eggs on satiety in overweight and obese subjects. J Am Coll Nutr. 2005 Dec;24(6):510-5. doi: 10.1080/07315724.2005.10719497. PMID 16373948